CLINICAL TRIAL: NCT00782054
Title: Evaluation of Provase in the Post Burn Rehabilitation Population for Itch Control and Moisturization Properties
Brief Title: Evaluation of Post Burn Rehabilitation Population for Itch Control
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Swiss-American Products, Inc (Industry)
Collaborators: McGill University (Other); Hospital de readaptation Villa Medica (Unknown); Precision Consulting (Unknown)
Responsible Party: Leo LaSalle, Hospital de readaptation Villa Medica
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-05-08573
Record Dates: First submitted 2008-10-27; First posted 2008-10-29 (Estimated); Last update posted 2008-10-29 (Estimated); Status verified 2008-10

CONDITIONS: Pruritus; Itching; Burn Pruritus
Keywords: pruritus; itch; burn; endopeptidase; moisturizer; randomized controlled
MeSH Terms: conditions — Pruritus; Burns

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Active Comparator): moisturizer with endopeptidases
  Interventions: Other: Provase
- Placebo (Placebo Comparator): moisturizer without endopeptidases
  Interventions: Other: Control moisturizer

INTERVENTIONS:
Other: Provase — NDC:60230-8573-0 Over the counter (OTC) moisturizer containing 2% dimethicone and a blend of endopeptidases. Use topically to affected area every 8 hours.
  Arms: Active
Other: Control moisturizer — Over the counter (OTC) moisturizer containing 2% dimethicone. Use topically to affected area every 8 hours. Does NOT contain endopeptidases. Placebo intervention is identical to active intervention EXCEPT it does not contain endopeptidases.
  Arms: Placebo

SUMMARY:
Severe itching following burn injury is a common complication. As many as 87% of burn patients report severe itching. The intense itching can increase anxiety and can interfere with sleep and normal activities of daily living thus affecting quality of life. Often the itching will become so intense patients will scratch or rub the skin until an open wound develops. Current treatment for itching includes antihistamines, steroids. and/or moisturizers, but too often, the patient does not receive relief, even from drugs, and suffers undesirable side effects.

Swiss-American Products, Inc, has developed a new skin moisturizer containing a blend of endopeptidase enzymes. These products have resolved itching in other types of skin disease such as dermatitis. The hypothesis that itching can be reduced through the use of these endopeptidase enzyme containing products in the post burn population will be tested.

DETAILED DESCRIPTION:
The mechanism of pruritus is poorly understood, but much stems from the inflammatory process during wound healing. Damaged nerve endings, substance P, mast cells releasing histamines, and presence of inflammatory prostaglandins can induce neuropathic and peripheral pruritoceptive itching. Absence of oil glands leading to dry skin and itching further aggravate the itching.

Swiss-American Products, Inc, has developed new non-prescription skin products containing a blend of endopeptidase enzymes in a moisturizer base to aid the body during recovery from injury and inflammation. In Stage II and III pressure ulcers, an amorphous hydrogel containing the enzymes was observed to help resolve inflammation and enhance healing. Anecdotal reports indicate a fast release cream with the enzymes, applied to insect stings and bites on intact skin resolved the itching and reduced, sometimes even preventing, edema. In a case study of chronic persistent contact dermatitis, one product was successfully used for immediate relief of pruritus and the slow release version was used for relief at night. Several centers have independently reported the resolution of pruritus associated with cellulitis in subjects with chronic wounds.

The hypothesis that itching can be reduced through the use of endopeptidase enzyme containing product in the post burn population will be tested. The use of the product has not been previously evaluated in burn subjects with pruritus. The primary objective of the preliminarily study would be to detect reduction of post burn itching through the use of the endopeptidase enzyme containing product.

ELIGIBILITY:
Inclusion Criteria:

* Post burn subject must be experiencing pruritus as defined by
* at least three episodes of itch during the past week AND
* itching occurs at least twice during the episode day AND
* itching lasts for more than 5 minutes and is bothersome
* TBSA of burn is between 10 and 70%
* Currently performing rehabilitation at Villa Medica Rehabilitation Hospital
* Subject available for 4 weeks
* Test area has complete epithelialization
* Subject is willing to complete daily diary
* Subject is male or female and over 18 years of age

Exclusion Criteria:

* Subject will be excluded if pruritus is of nonburn etiology
* Subject requires topical steroids, topical antihistamines, or other topical medication and such medication cannot be discontinued
* Subject with known sensitivity to the enzyme papain or to the papaya fruit
* Subject requires immunosuppressives such as systemic steroid therapy, cancer chemotherapeutic agents
* Subject presently requires morphine for pain relief
* Subject is a known alcohol or drug abuser
* Subject is unable to communicate pain and itch scores or medication used

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-09; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
The primary variables will be the responses on the Yosipovitch and Matheson instruments for each sensation/affect of itch category (tickling, stinging, crawling, stabbing, pinching, burning) and on severity (none, mild, moderate, and severe). | 4 weeks

SECONDARY OUTCOMES:
Secondary variables include antihistamine usage, skin condition, scar evaluation, and subject acceptance. Safety will be assessed via collection of adverse events. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Leo LaSalle, M.D., Principal Investigator — Villa Medica Rehabilitation Hospital; Bernadette Nedelec, BSc, OT, PhD, Study Chair — McGill University
Locations (1):
- Villa Medica Rehabilitation Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] Field T, Peck M, Scd, Hernandez-Reif M, Krugman S, Burman I, Ozment-Schenck L. Postburn itching, pain, and psychological symptoms are reduced with massage therapy. J Burn Care Rehabil. 2000 May-Jun;21(3):189-93. doi: 10.1067/mbc.2000.105087. PMID 10850898
- [Background] Dunnick CA, Gibran NS, Heimbach DM. Substance P has a role in neurogenic mediation of human burn wound healing. J Burn Care Rehabil. 1996 Sep-Oct;17(5):390-6. doi: 10.1097/00004630-199609000-00004. PMID 8889861
- [Background] Yosipovitch G, Fleischer A. Itch associated with skin disease: advances in pathophysiology and emerging therapies. Am J Clin Dermatol. 2003;4(9):617-22. doi: 10.2165/00128071-200304090-00004. PMID 12926980
- [Background] Matheson JD, Clayton J, Muller MJ. The reduction of itch during burn wound healing. J Burn Care Rehabil. 2001 Jan-Feb;22(1):76-81; discussion 75. doi: 10.1097/00004630-200101000-00017. PMID 11227690
- [Background] Baker RA, Zeller RA, Klein RL, Thornton RJ, Shuber JH, Marshall RE, Leibfarth AG, Latko JA. Burn wound itch control using H1 and H2 antagonists. J Burn Care Rehabil. 2001 Jul-Aug;22(4):263-8. doi: 10.1097/00004630-200107000-00003. PMID 11482684
- [Background] Parnell LK, Ciufi B, Gokoo CF. Preliminary use of a hydrogel containing enzymes in the treatment of stage II and stage III pressure ulcers. Ostomy Wound Manage. 2005 Aug;51(8):50-60. PMID 16234576
- [Background] Barnett L, Parnell LK. Contact dermatitis treated with new topical products: a case study. Ostomy Wound Manage. 2001 Sep;47(9):47-53. PMID 11889744
- [Background] Yosipovitch G, Goon AT, Wee J, Chan YH, Zucker I, Goh CL. Itch characteristics in Chinese patients with atopic dermatitis using a new questionnaire for the assessment of pruritus. Int J Dermatol. 2002 Apr;41(4):212-6. doi: 10.1046/j.1365-4362.2002.01460.x. PMID 12031029
- [Background] Yosipovitch G, Zucker I, Boner G, Gafter U, Shapira Y, David M. A questionnaire for the assessment of pruritus: validation in uremic patients. Acta Derm Venereol. 2001 May;81(2):108-11. doi: 10.1080/00015550152384236. PMID 11501646
- [Background] Nedelec B, Shankowsky HA, Tredget EE. Rating the resolving hypertrophic scar: comparison of the Vancouver Scar Scale and scar volume. J Burn Care Rehabil. 2000 May-Jun;21(3):205-12. doi: 10.1067/mbc.2000.104750. PMID 10850901
- See also: McGill University Homepage — http://www.mcgill.ca
- See also: Villa Medica Rehabilitation Hospital Homepage — http://www.villamedica.ca